CLINICAL TRIAL: NCT02208596
Title: The Feasibility of Different Doses of Etomidate Admixed With Propofol in Induced Abortion: A Randomized, Double Blind Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140729
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Induced Abortion; Anesthesia
MeSH Terms: interventions — Pentazocine; Propofol; Etomidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): In group A, propofol (1%) was mixed with etomidate in the ration of 1:1 (volume). The mixture will be injected continuously until the eyelash reflex disappears. During the operation, supplementary mixture will be administered if the patient has spontaneous movement that hampered the conduct of the procedure.
  Interventions: Drug: pentazocine; Drug: propofol; Drug: Etomidate
- Group B (Experimental): In group B, propofol (1%) was mixed with etomidate in the ration of 7:5 (volume). The mixture will be injected continuously until the eyelash reflex disappears. During the operation, supplementary mixture will be administered if the patient has spontaneous movement that hampered the conduct of the procedure.
  Interventions: Drug: pentazocine; Drug: propofol; Drug: Etomidate
- Group C (Experimental): In group C, propofol (1%) will be injected continuously until the eyelash reflex disappears. During the operation, supplementary propofol will be administered if the patient has spontaneous movement that hampered the conduct of the procedure.
  Interventions: Drug: pentazocine; Drug: propofol

INTERVENTIONS:
Drug: pentazocine — Every patient enrolled in the study will be given 15 mg pentazocine before induction.
Drug: propofol
Drug: Etomidate
  Arms: Group A; Group B

SUMMARY:
To explore the feasibility of different doses of etomidate admixed with propofol in induced abortion: a randomized, double blind controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 35 years
* American Society of Anesthesiology (ASA) Physical Status: Ⅰ or Ⅱ
* Singleton pregnancy and the gestational period is 6 to 8 weeks
* Expected operation duration is within 60 minutes
* The body weight should be within 15% around the standard weight
* Signed informed consent form

Exclusion Criteria:

* Serious cardiac, cerebral, liver, kidney, lung, endocrine disease
* Upper respiratory infections within 4 weeks
* Long use of hormone or history of adrenal suppression
* History of use of glucocorticoids, aprotinin or immunosuppressant
* Manifestation of immunodeficiency
* History of use of sedatives or opiates
* Needs of Neuromuscular blocker (except intubation)
* Allergy to trial drug or other contraindication
* Pregnant or breast-feeding women
* Attended other trial past 30 days

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Heart rate | From baseline (before the injection of propofol or mixture of propofol and etomidate) to 10 min after the injection
  Heart rate will be recorded immediately when the patient arrived at the operating room, 2 min, 4 min, 6 min, 8 min and 10 minutes after the the injection of propofol or mixture of propofol and etomidate.
Blood pressure | From baseline (before the injection of propofol or mixture of propofol and etomidate) to 10 min after the injection
  Blood pressure will be recorded immediately when the patient arrived at the operating room, 2 min, 4 min, 6 min, 8 min and 10 minutes after the the injection of propofol or mixture of propofol and etomidate.
Pulse oxygen saturation | From baseline (before the injection of propofol or mixture of propofol and etomidate) to 10 min after the injection
  Pulse oxygen saturation will be recorded immediately when the patient arrived at the operating room, 2 min, 4 min, 6 min, 8 min and 10 minutes after the the injection of propofol or mixture of propofol and etomidate.

SECONDARY OUTCOMES:
Efficacy of anesthesia | from baseline to discharge from the hospital, expected to no more than 1 hour
  The following point-in-time will be recorded to calculated the period from the injection of propofol or mixture of propofol and etomidate: disappearance of eyelash reflex, injection of supplementary propofol or mixture of propofol and etomidate, awaking, obeying commands, discharge. Anesthesia time was defined as the period from disappearance of eyelash reflex to awaking.
Dose of propofol or mixture of propofol and etomidate | from the injection of propofol or mixture of propofol and etomidate to the last supplement of hypnotic agents, expected to be no more than 5 min
Use of specific medications | from the injection of propofol or mixture of propofol and etomidte to discharge from the hospital, expected to no more than 1 hour
Aldrete score | 10 min after the opration
Verbal rating scales of uterine contraction | from 5 min after the operation to discharge from the hospital, expected to be no more than 1 hour
  Verbal rating scales of uterine contraction should be recorded at 5 min, 15 min after the operation and before discharge from the hospital
Satisfaction degree of the patient, the surgeon and the anesthetist | 10 min before discharge from the hospital
  Satisfaction degree will be rated as excellent, good and poor based on a scale of 1 to 10. Excellent is 8 to 10, good is 5 to 7 and poor is 1 to 4.